CLINICAL TRIAL: NCT06909747
Title: The Effects of Posture Training Given to Middle School Students on Back Pain and Body Posture: A Randomized Controlled Study
Brief Title: Posture Training for Middle Schoolers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Aslı Yılmaz, Vice Dean of Faculty of Health Sciences, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025000051
Record Dates: First submitted 2025-03-26; First posted 2025-04-03 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-03

CONDITIONS: Musculoskeletal Pain; Postural; Defect
Keywords: body posture; back pain; mid-school student; health education
MeSH Terms: conditions — Musculoskeletal Pain; Back Pain; Health Education

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): The experimental group will be given training planned in a total of three sessions on correct body posture and spinal health and its importance, and exercises to be done for spinal health.
  Interventions: Behavioral: Posture Training
- Control Group (No Intervention): No intervention will be applied.

INTERVENTIONS:
Behavioral: Posture Training — Training program consists of three sessions. It will cover proper body posture, the importance of spinal health, and targeted exercises to support spinal well-being.
  Arms: Training Group

SUMMARY:
The goal of this clinical trial is to investigate if posture training can improve back pain and posture in middle school students. The main questions it aims to answer are:

* Can posture training reduce back pain in middle school students?
* Can posture training improve body posture in middle school students?

Researchers will compare training and control groups to see if posture training reduces pain and improves body posture.

Participants will;

* Fill a survey assessing pain and body posture at three time points: before the training, immediately after, and at the 1st and 3rd months
* Attend three sessions of training on correct body posture and spinal health and its importance, and exercises to be done for spinal health

DETAILED DESCRIPTION:
This experimental study has been designed with a pre-test-post-test control group and repeated-measures. The data will be collected between October 15, 2025 and March 15, 2026. The study will be conducted in two Middle School in a region with a total students of 1170 in the 2024-2025 academic year. It is assumed that the population size will be similar, and a power analysis (0.80 power and 0.05 margin of error) has been conducted to estimate the sample size. As a result the target is to reach a total of 80 students, with 40 students in both the experimental and control groups, including a 20% attrition rate. The study will begin after the institutional permission, ethics committee approval, and written consent from the parents and verbal consent from the students. After the pre-test is completed, the students in the experimental group will be given training planned in a total of three sessions on correct body posture and spinal health and its importance, and exercises to be done for spinal health. The research data will be collected before and after the intervention, in the 1st and 3rd months. In the study, the data will be collected with the personal information form prepared by the researchers in line with the literature information and the Back Pain and Body Posture Assessment Tool, the validity and reliability of which has been studied in Turkish. In this study, the Statistical Package for Social Science for Windows (SPSS) package program will be used to analyse, examine and perform the analysis of the data.

In the data analysis, ordinal variables will be evaluated as arithmetic mean and standard deviation, minimum, maximum. As statistical analysis methods, Student's t test and one-way variance (One Way ANOVA), and Mann-Whitney U test will be used, and the significance level will be considered at p<0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent and voluntary participation
* No physical or mental disabilities
* Being a 5th, 6th, 7th, or 8th-grade student
* Marking inappropriate posture (incorrect answer) in at least 4 out of 5 posture-related questions in the Back Pain and Posture Assessment tool
* Being present at school on the study days, with no excused absence or medical leave
* Full participation in the training program and completion of the follow-up process after the pre-test

Exclusion Criteria:

* Lack of parental consent
* Voluntary withdrawal from the study
* Failure to complete all three training sessions
* Inability to attend school for any reason
* Presence of a chronic condition that may cause back pain or posture disorders

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Back pain | Baseline, Month 1 and Month 3
  This will be assessed with a validated tool called Back Pain and Body Posture Assessment Tool
Body Posture | Baseline, Month 1 and Month 3
  This will be assessed with a validated tool called Back Pain and Body Posture Assessment Tool

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Yılmaz, Dr, Principal Investigator — Vice Dean of Faculty of Health Sciences
Locations (2):
- Turkey (Türkiye) (2):
  - Amasya Serdar Zeren Middle School, Amasya
  - Amasya Yavuz Selim Middle School, Amasya

IPD SHARING:
Plan to Share IPD: No